CLINICAL TRIAL: NCT05477277
Title: Adverse Outcomes and Mortality in Liver Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Amra Medical AB (Industry)
Responsible Party: Principal Investigator, Elizabeth Carey, Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-007442
Record Dates: First submitted 2022-07-12; First posted 2022-07-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: End Stage Liver DIsease; Sarcopenia; Sarcopenic Obesity; Cirrhosis
MeSH Terms: conditions — End Stage Liver Disease; Sarcopenia; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Define MAsS cut-point at transplant evaluation to identify those with high risk for adverse outcomes (Experimental)
  Interventions: Diagnostic Test: MAsS

INTERVENTIONS:
Diagnostic Test: MAsS — Add MAsS to standard of care MRI scan

SUMMARY:
Prospective natural history pilot study to explore the link between muscle composition using an MRI-based Muscle Assessment Score (MAsS) and adverse outcomes in liver transplant candidates.

DETAILED DESCRIPTION:
Sarcopenia, characterized by the progressive loss of muscle volume and function, is a common and major complication in end-stage liver disease which significantly contributes to adverse outcomes and mortality as well as hampers successful outcomes for treatments such as liver transplant (LT). High resolution image-based techniques have been instrumental in furthering our understanding of body composition in sarcopenia specifically and human health in general. While several methods exist to evaluate body composition, imaging techniques, such as computed tomography (CT) and magnetic resonance imaging (MRI) enable capitalization of images taken as part of standard practice as well as append already clinical examinations with brief sequences tailored for mapping muscle and body composition. Opportunistic application of this imaging-based body composition assessment to patients in a liver transplant context has revealed a high prevalence of sarcopenia (low muscle volume relative to age and sex) and pathological muscle fat infiltration (myosteatosis). Furthermore, a recent long-term (6-years post-LT) MRI-based retrospective study showed associations of myosteatosis to increased graft loss and mortality after transplant.

The combination of MRI-based thigh muscle volume and fat infiltration has been suggested as a more complete description of muscle composition with a stronger link to hospitalization, poor functional activities of daily life, and metabolic co-morbidities in general population and subjects presenting with non-alcoholic fatty liver disease. A recently submit paper explored the predictive power of this combination based on 40 000 participants in the UK biobank and found that the presence of adverse muscle composition, that is the combination of lower-than-expected muscle volume and high muscle fat infiltration, showed to be a strong and independent predictor of all-cause mortality comparable to that of previous cancer diagnosis and smoking. The same MRI-sequence and body composition assessment has successfully been implemented in small pilot studies before and after LT, both within weeks and years after LT, and presented at recent scientific conferences.

There is a lack of knowledge in how to fully identity patients indicted for liver transplant that are of very high risk for adverse outcomes and mortality in standardized fashion. The aim is to use an MRI-based Muscle Assessment Score (MAsS), which includes both muscle volume and fat infiltration, at the transplant candidacy evaluation and other follow-up MRI examinations as clinically indicated, as an objective, standardized, and quantitative measure of muscle health and explore the link between muscle composition and adverse outcomes and mortality. In addition, there are growing numbers of high-risk donor livers, such as presenting with steatosis or exposed to prolonged ischemia time. A co-primary aim is to gather information on the association between transplant recipient muscle composition and donor liver characteristics to one-year post-LT adverse outcomes and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with end-stage liver disease undergoing evaluation for liver transplantation
2. Patient clinically indicated for MRI during transplant candidacy evaluation
3. Adult

Exclusion Criteria:

1. Contra indication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Muscle assessment score (MAsS) | 1 year
  The MAsS is a composite score of muscle fat index (% of muscle fat normalized to sex, weight in kg and height in meters) and muscle volume index (muscle volume in liters normalized to patient sex, height in meters and weight in kg)
Adverse outcomes | 1 year
  Number of pre- and post-transplant inpatient days
Adverse outcomes | 1 year
  Number of pre- and post-transplant ICU days
Adverse outcomes | 1 year
  Number of days alive outside of the hospital in the first year after liver transplant
Adverse outcomes | 1 year
  Mortality within the first year after liver transplant
MAsS changes while waiting for liver transplant | 1 year
  In patients who remain on the waitlist, serial MAsS measurements (see Outcome 1) will be taken and changes over time will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Elizabet Carey, MD, Principal Investigator — Mayo Cinic
Locations (1):
- Mayo Clinic Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borga M, Thomas EL, Romu T, Rosander J, Fitzpatrick J, Dahlqvist Leinhard O, Bell JD. Validation of a fast method for quantification of intra-abdominal and subcutaneous adipose tissue for large-scale human studies. NMR Biomed. 2015 Dec;28(12):1747-53. doi: 10.1002/nbm.3432. Epub 2015 Nov 2. PMID 26768490
- [Background] Borga M, West J, Bell JD, Harvey NC, Romu T, Heymsfield SB, Dahlqvist Leinhard O. Advanced body composition assessment: from body mass index to body composition profiling. J Investig Med. 2018 Jun;66(5):1-9. doi: 10.1136/jim-2018-000722. Epub 2018 Mar 25. PMID 29581385
- [Background] Carey EJ, Lai JC, Sonnenday C, Tapper EB, Tandon P, Duarte-Rojo A, Dunn MA, Tsien C, Kallwitz ER, Ng V, Dasarathy S, Kappus M, Bashir MR, Montano-Loza AJ. A North American Expert Opinion Statement on Sarcopenia in Liver Transplantation. Hepatology. 2019 Nov;70(5):1816-1829. doi: 10.1002/hep.30828. Epub 2019 Aug 19. PMID 31220351
- [Background] Feng S, Goodrich NP, Bragg-Gresham JL, Dykstra DM, Punch JD, DebRoy MA, Greenstein SM, Merion RM. Characteristics associated with liver graft failure: the concept of a donor risk index. Am J Transplant. 2006 Apr;6(4):783-90. doi: 10.1111/j.1600-6143.2006.01242.x. PMID 16539636
- [Background] Flores A, Asrani SK. The donor risk index: A decade of experience. Liver Transpl. 2017 Sep;23(9):1216-1225. doi: 10.1002/lt.24799. PMID 28590542
- [Background] Karlsson A, Rosander J, Romu T, Tallberg J, Gronqvist A, Borga M, Dahlqvist Leinhard O. Automatic and quantitative assessment of regional muscle volume by multi-atlas segmentation using whole-body water-fat MRI. J Magn Reson Imaging. 2015 Jun;41(6):1558-69. doi: 10.1002/jmri.24726. Epub 2014 Aug 11. PMID 25111561
- [Background] Linge J, Borga M, West J, Tuthill T, Miller MR, Dumitriu A, Thomas EL, Romu T, Tunon P, Bell JD, Dahlqvist Leinhard O. Body Composition Profiling in the UK Biobank Imaging Study. Obesity (Silver Spring). 2018 Nov;26(11):1785-1795. doi: 10.1002/oby.22210. Epub 2018 May 22. PMID 29785727
- [Background] Linge J, Heymsfield SB, Dahlqvist Leinhard O. On the Definition of Sarcopenia in the Presence of Aging and Obesity-Initial Results from UK Biobank. J Gerontol A Biol Sci Med Sci. 2020 Jun 18;75(7):1309-1316. doi: 10.1093/gerona/glz229. PMID 31642894
- [Background] Linge J, Ekstedt M, Dahlqvist Leinhard O. Adverse muscle composition is linked to poor functional performance and metabolic comorbidities in NAFLD. JHEP Rep. 2020 Oct 28;3(1):100197. doi: 10.1016/j.jhepr.2020.100197. eCollection 2021 Feb. PMID 33598647
- [Background] Linge J, Petersson M, Forsgren MF, Sanyal AJ, Dahlqvist Leinhard O. Adverse muscle composition predicts all-cause mortality in the UK Biobank imaging study. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1513-1526. doi: 10.1002/jcsm.12834. Epub 2021 Oct 29. PMID 34713982
- [Background] Montano-Loza AJ, Angulo P, Meza-Junco J, Prado CM, Sawyer MB, Beaumont C, Esfandiari N, Ma M, Baracos VE. Sarcopenic obesity and myosteatosis are associated with higher mortality in patients with cirrhosis. J Cachexia Sarcopenia Muscle. 2016 May;7(2):126-35. doi: 10.1002/jcsm.12039. Epub 2015 Jun 9. PMID 27493866
- [Background] Shenvi SD, Taber DJ, Hardie AD, Botstein JO, McGillicuddy JW. Assessment of magnetic resonance imaging derived fat fraction as a sensitive and reliable predictor of myosteatosis in liver transplant recipients. HPB (Oxford). 2020 Jan;22(1):102-108. doi: 10.1016/j.hpb.2019.06.006. Epub 2019 Aug 9. PMID 31405777
- [Background] West J, Dahlqvist Leinhard O, Romu T, Collins R, Garratt S, Bell JD, Borga M, Thomas L. Feasibility of MR-Based Body Composition Analysis in Large Scale Population Studies. PLoS One. 2016 Sep 23;11(9):e0163332. doi: 10.1371/journal.pone.0163332. eCollection 2016. PMID 27662190
- [Background] West J, Romu T, Thorell S, Lindblom H, Berin E, Holm AS, Astrand LL, Karlsson A, Borga M, Hammar M, Leinhard OD. Precision of MRI-based body composition measurements of postmenopausal women. PLoS One. 2018 Feb 7;13(2):e0192495. doi: 10.1371/journal.pone.0192495. eCollection 2018. PMID 29415060